CLINICAL TRIAL: NCT00000304
Title: Dextroamphetamine as an Adjunct in Cocaine Treatment
Brief Title: Dextroamphetamine as an Adjunct in Cocaine Treatment - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Texas (Other)
Responsible Party: F.Gerard Moeller, University of Texas Medical School at Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-09262-1; P50-09262-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Cocaine-Related Disorders; Substance-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Dextroamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 15/30 mg d-amphetamine
  Interventions: Drug: Dextroamphetamine
- 2 (Experimental): 30/60 mg d-amphetamine
  Interventions: Drug: D-Amphetamine
- 3 (Experimental): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dextroamphetamine — 15 mg for first 8 weeks and 30 mg for 2nd 8 weeks
  Arms: 1
Drug: D-Amphetamine — 30 mg for the first 8 weeks and 60 for the second 8 weeks (16 weeks total)
  Arms: 2
Drug: Placebo — Placebo
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate dextroamphetamine sulfate (sustained release) as an adjunct in cocaine treatment; an evaluation of the ""replacement"" strategy.

ELIGIBILITY:
Please contact site for information.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 1997-08; Primary Completion 2001-08 (Actual); Study Completion 2001-08 (Actual)

PRIMARY OUTCOMES:
verifiable cocaine abstinence | 16 weeks of study

CONTACTS AND LOCATIONS:
Overall Officials: John Grabowski, Ph.D., Principal Investigator — University of Texas
Locations (1):
- University of Texas Health Science Center, Houston, Texas, United States